CLINICAL TRIAL: NCT04423861
Title: A Phase III, Multicentre, Parallel, Randomized, Double-blind Clinical Trial to Assess the Efficacy and Safety of Nitazoxanide 600 mg Compared to Placebo in the Treatment of Hospitalized Patients With COVID-19 in Non-critical Condition
Brief Title: Efficacy and Safety of Nitazoxanide 600 mg BID Versus Placebo for the Treatment of Hospitalized Patients With COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azidus Brasil (Industry)
Collaborators: Farmoquimica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NITFQM0920OR-III
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: covid19
MeSH Terms: conditions — COVID-19 | interventions — nitazoxanide

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either nitazoxanide 600 mg BID or Placebo (1:1)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nitazoxanide BID (Experimental): Patients will receive nitazoxanide 600 mg BID for 7 days.
  Interventions: Drug: Nitazoxanide
- Placebo (Placebo Comparator): Patients will receive matching placebo BID for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitazoxanide — Patients will receive nitazoxanide 600 mg BID for 7 days.
  Other Names: Viranitta (Nitazoxanide)
  Arms: nitazoxanide BID
Drug: Placebo — Patients will receive matching placebo BID for 7 days.
  Arms: Placebo

SUMMARY:
This is a pivotal phase III study to evaluate the efficacy of nitazoxanide 600 mg BID compared to placebo to treat hospitalized patients with non-critical COVID-19.

DETAILED DESCRIPTION:
This is pivotal phase III study to evaluate the efficacy of nitazoxanide 600 mg BID compared to placebo to treat hospitalized patients with non-critical COVID-19.

The aim is to demonstrate a decrease in hospital related complications among patients who are hospitalized with moderate COVID-19 by treating them with nitazoxanide BID 600 mg for 7 days on top of standard care compared to placebo on top of standar care..

Therefore, patients hospitalized with confirmed diagnosis of COVID-19 will be randomized to receive either nitazoxanide 600 mg BID or Placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent from patient or legal representative.
2. Male or female, aged ≥ 18 years;
3. Laboratory confirmation of 2019-nCoV infection by reverse-transcription polymerase
4. chain reaction (RT-PCR) from any diagnostic sampling source;
5. Hospitalized for up to 48h with signs of respiratory failure with or without non-invasive ventilation and i. Oxygen saturation <98%;

7. Negative result for pregnancy test (if applicable).

Exclusion Criteria:

1. Participating in another RCT in the past 12 months;
2. Known allergy to nitazoxanide
3. Severely reduced LV function;
4. Severely reduced renal function;
5. Pregnancy or breast feeding;
6. Diagnosis of any other active infection (viral, bacterial, fungal or caused by another pathogen, except the one studied in the trial);
7. History of HIV 1 and/or 2 (Anti-HIV-1,2) and/or HTLV I and II positive;
8. Ongoing antineoplastic treatment with chemotherapy or radiation therapy;
9. Diagnose of severe autoimmune diseases in immunosuppression;
10. Transplanted patients;
11. Any other clinical condition which, in the opinion of the principal investigator, would not allow safe completion of the protocol and safe administration of the investigational products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Need of mechanical ventilation | 14 days
  Evaluation of change in acute respiratory syndrome using WHO Ordinal Scale for Clinical Improvement that measures illness severity over time (0=uninfected; ambulatory, no limitation of activities=1; ambulatory, limitation of activities=2, hospitalized no oxygen therapy=3; hospitalized oxygen by mask or nasal prongs=4; hospitalized non invasive ventilation or high-flow oxygen=5; hospitalized intubation or mechanical ventilation=6; hospitalized ventilation + additional organ support=7; death=8)

SECONDARY OUTCOMES:
Change in the pulmonary condition | Baseline, Day 7 and Day 14
  Evaluation of change in oximetry, respiratory rate and need for oxygen therapy
Change in Clinical Condition | Baseline, Day 7 and Day 14
  Evaluation of change in the following symptoms: cough, headache, myalgia and fever, level of consciousness and organ dysfunction
Change in tomographic pulmonary condition | Baseline, Day 7
  Evaluation of change in chest CT
Rate of mortality within 14-days | 14 days
  Evaluation of change in acute respiratory syndrome
Change in inflammatory markers | Baseine, Day 7, Day 14
  Evaluation of change in inflammatory markers d-dimer and IL-6

CONTACTS AND LOCATIONS:
Overall Officials: Florentino de Araujo Cardoso Filho, MD, PhD, Principal Investigator — +55 19 991232882
Locations (1):
- Hospital Vera Cruz, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
It is believed that after the data analysis and presentation to the National Commission on Research Ethics, all data of the study will become public.